CLINICAL TRIAL: NCT06831903
Title: Simultaneous Integrated Boost in the Primary and Adjuvant Therapy of Head and Neck Cancer: Quality Control Registry Prospective Longitudinal Obervation Trial
Brief Title: Radiotherapy of Head and Neck Cancer With SIB
Status: Recruiting | Type: Observational
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 159/16-sc
Record Dates: First submitted 2025-01-03; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Quality of Life (QOL); Head and Neck Cancer; Radiotherapy Side Effect; Radiotherapy, Conformal (IMRT)
MeSH Terms: conditions — Head and Neck Neoplasms; Radiation Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Head and neck radio(chemo)therapy: Patients aged 18 and older with histologically confirmed malignant head and neck tumors, undergoing definitive or adjuvant radio(chemo)therapy at the University Hospital Würzburg between October 2019 and October 2034.

SUMMARY:
Title: Simultaneous Integrated Boost in Primary and Adjuvant Therapy of Head and Neck Tumors: Quality Control Registry Prospective Longitudinal Observational Study

Short Title: Radiotherapy for Head and Neck Tumors with SIB

Objective: To evaluate the efficacy and safety of definitive and adjuvant radio(chemo)therapy with simultaneous integrated boost (SIB) in patients with head and neck cancers. The study aims to assess local and regional control, overall survival, metastasis-free survival, therapy-related toxicities, and quality of life.

Study Design: A prospective, longitudinal, non-interventional registry study documenting real-world outcomes and quality measures of therapy applied according to existing clinical guidelines.

DETAILED DESCRIPTION:
This study is a prospective, longitudinal, non-interventional quality control registry focused on the application of simultaneous integrated boost intensity-modulated radiotherapy (SIB-IMRT) in the primary and adjuvant treatment of head and neck cancers. The primary objectives are to evaluate local and regional control rates, overall survival, tumor-specific survival, and metastasis-free survival. The study also aims to document acute and late treatment-associated toxicities, patient-reported quality of life, and recurrence patterns in relation to delivered radiation doses.

Patients with histologically confirmed malignancies of the head and neck region (excluding basal cell carcinoma) who are indicated for definitive or adjuvant radiotherapy or radiochemotherapy will be included. Treatment planning involves individualized IMRT/VMAT-based approaches with SIB techniques designed to escalate doses to high-risk tumor regions while sparing surrounding healthy structures, thereby reducing toxicity. The treatment is provided in compliance with national guidelines and inter-disciplinary tumor board recommendations.

Evaluation of Adverse Events The study employs the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaires-QLQ-C30 and H&N35-to systematically assess treatment-related adverse events (AEs) and their impact on quality of life. These standardized tools are administered at baseline, at the end of treatment, and during follow-up visits.

The EORTC QLQ-H&N35 questionnaire, specifically tailored for head and neck cancer patients, captures detailed information on a wide range of symptoms and treatment-related toxicities, including but not limited to:

Swallowing and Oral Function:

Dysphagia (difficulty swallowing) Speech problems (articulation and clarity) Xerostomia (dry mouth) Sticky saliva

Sensory Impairments:

Altered taste and smell Hearing loss

Pain and Discomfort:

Pain in the mouth, throat, or jaw Soreness or discomfort in the treated area

Respiratory Symptoms:

Breathing difficulties Nasal congestion or discharge

Nutritional Challenges:

Difficulty eating or maintaining weight Nutritional supplementation requirements

Emotional and Social Impact:

Body image concerns Social functioning and isolation Financial burden associated with treatment

Other Common Toxicities:

Skin reactions in the irradiated area Fatigue and general physical discomfort These adverse events are graded using the Common Terminology Criteria for Adverse Events (CTCAE), enabling consistent reporting of the severity and frequency of toxicities.

Data Collection and Statistical Analysis The collected data will include baseline patient characteristics, treatment parameters, and longitudinal quality-of-life scores. Outcomes will be analyzed to identify correlations between reported toxicities, dosimetric parameters, and clinical outcomes, such as recurrence patterns and survival metrics.

The statistical methodology includes:

Descriptive statistics for baseline demographics and treatment variables. Kaplan-Meier estimates for survival analysis. Cox proportional hazards models to explore the influence of clinical and treatment-related factors on survival and recurrence.

Correlation analyses to assess the relationship between dosimetric variables and recurrence patterns.

Significance of the Study This study seeks to complement clinical trial data with real-world evidence on the implementation of SIB-IMRT in head and neck cancer treatment. By systematically capturing and analyzing treatment-related toxicities and quality-of-life metrics, the findings aim to refine therapeutic protocols, enhance patient outcomes, and inform strategies to mitigate adverse events. Moreover, the integration of recurrence pattern analysis and ontogenetic lymphatic mapping could offer valuable insights for future treatment planning.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and older with histologically confirmed malignant head and neck tumors, undergoing definitive or adjuvant radio(chemo)therapy at the University Hospital Würzburg

Exclusion Criteria:

* missing informed consent
* mental or physical disorders leading to inability to understand and/or fill the quationary
* judgment by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 and older with histologically confirmed malignant head and neck tumors, undergoing definitive or adjuvant radio(chemo)therapy at the University Hospital Würzburg between October 2019 and October 2034
Sampling Method: Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2019-05-21 (Actual); Primary Completion 2034-10-01 (Estimated); Study Completion 2039-10-01 (Estimated)

PRIMARY OUTCOMES:
Local control rate. | From the date of treatment initiation until local recurrence or last follow-up, whichever occurs first, assessed up to 60 months.
  Key aspects of local tumor control include:
  No Evidence of Tumor Growth:
  The absence of measurable or observable increase in the size of the tumor at the primary site.
  Tumor Response to Treatment:
  Complete Response (CR): Disappearance of all signs of cancer at the primary site.
  Partial Response (PR): Reduction in tumor size without complete disappearance.
  Persistence of Stable Disease:
  The tumor remains unchanged in size and does not spread locally beyond the treated area.
  Time Frame: 5 years from treatment start.
  Assessment Methods:
  Clinical Examination: Evaluation of the treated site for physical signs of recurrence.
  Imaging Techniques: CT, MRI, or PET scans to detect residual or recurrent disease.
  Biopsy: When clinically indicated, to confirm recurrence if suspected.
Regional tumor control rate | From the date of treatment initiation until regional recurrence or last follow-up, whichever occurs first, assessed up to 60 months.
  Key aspects of regional tumor control include:
  Absence of Disease Progression:
  No enlargement, growth, or new involvement of lymph nodes in the regional drainage area.
  Response to Treatment:
  Complete Response (CR): All detectable cancer in the regional lymph nodes has disappeared.
  Partial Response (PR): A significant reduction in the size of affected lymph nodes or nodal masses.
  Stable Disease:
  The size and characteristics of the regional lymph nodes remain unchanged after treatment, without evidence of further spread.
  Time Frame: 5 years
  Assessment Methods:
  Imaging: CT, MRI, or PET scans are used to assess lymph node involvement and detect residual or recurrent disease.
  Physical Examination: Palpation or clinical inspection for lymph node abnormalities.
  Biopsy or Fine Needle Aspiration: To confirm suspected recurrence or residual

SECONDARY OUTCOMES:
Overall Survival (OS) | From the date of treatment initiation until death from any cause or last follow-up, whichever occurs first, assessed up to 60 months.
  Overall Survival (OS) is a clinical endpoint that refers to the length of time from the start of treatment (or diagnosis, depending on the study design) until death from any cause.
  Key Aspects of Overall Survival:
  Inclusion of All Causes of Death:
  OS accounts for death from cancer, treatment-related complications, or any other unrelated causes (e.g., accidents or comorbid conditions).
  Measurement:
  OS as a median survival time (e.g., the time by which 50% of patients are still alive) and as a survival rate at specific time intervals (e.g., 1-year, 3 Year, 5-year OS rates).
  Time Frame:
  The starting point for measuring OS is the date of treatment initiation, The endpoint is the date of death or the last follow-up for patients who are still alive (censored data).
  Assessment Methods:
  OS is determined using survival analysis techniques, (Kaplan-Meier estimates), to calculate survival probabilities and generate survival curves.
Disease-Specific Survival (DSS) | From the date of treatment initiation until disease-specific death or last follow-up, whichever occurs first, assessed up to 60 months.
  Disease-Specific Survival (DSS) refers to the length of time from the start of treatment (or diagnosis, depending on the study design) until death specifically caused by the disease being studied, excluding deaths from other causes.
  Key Aspects of Disease-Specific Survival:
  Focus on Disease-Related Deaths:
  Only deaths directly attributable to the disease (e.g., cancer progression, metastasis) are considered in DSS calculations.
  Deaths from unrelated causes, such as accidents, other illnesses, or age-related factors, are excluded.
  Measurement:
  DSS is expressed as the time from treatment initiation to disease-specific death, or as a survival rate at specific intervals (e.g., 1,3,5-year DSS rate).
  Time Frame:
  The starting point for DSS measurement is the date of the start of treatment. The endpoint is the date of disease-specific death or last follow-up (for censored cases).
  Assessment Methods:
  DSS is determined using survival analysis techniques (Kaplan-Meier curves).
Metastasis-Free Survival (MFS) | From the date of treatment initiation until the first occurrence of distant metastasis, death from any cause, or last follow-up, whichever occurs first, assessed up to 60 months.
  MFS refers to the length of time from the start of treatment (or diagnosis, depending on the study design) until the first occurrence of distant metastasis (cancer spreading to distant organs or tissues) or death from any cause, whichever comes first. It is a commonly used endpoint in oncology studies to evaluate the effectiveness of treatments in preventing the spread of cancer.
  Inclusion Criteria:
  Patients are considered metastasis-free as long as there is no evidence of cancer spreading beyond the primary site and regional lymph nodes.
  Events Considered:
  Development of distant metastases (e.g. cancer in the lungs, liver, bones, or other remote organs).
  Death from any cause will be included in MFS, making it a composite endpoint.
  Measurement:
  MFS is expressed as the time from diagnosis or treatment initiation to the occurrence of distant metastasis or death. For patients who remain alive and free of metastases at the end of follow up the data are censored at the last FU.
Secondary malignancies | From Enrollment to the 5 years after the end of treatment.
  Incidence of secondary malignancies
Toxicities | From the date of enrollment until the occurrence of acute or late therapy-related toxicities, death, or last follow-up, whichever occurs first, assessed up to 60 months.
  Acute and late therapy-related toxicities (CTC AE scale).
General quality of life (EORTC QLQ-30) | Enrollment, end of radiotherapy (week 7 from start), week 6-8 after the end of radiotherapy, 12, 24, 36, 48, 60 Month after the end of radiotherapy or death from any cause, or last follow-up, whichever occurs first.
  The EORTC QLQ-C30 is a validated tool comprising 30 items grouped into functional scales (e.g., physical, emotional, and social functioning), symptom scales (e.g., fatigue, nausea, and pain), and global health status/QoL. Scores for each scale range from 0 to 100. Higher scores on functional and global health/QoL scales indicate better outcomes, whereas higher scores on symptom scales represent worse outcomes.
Organ specific quality of life (EORTC QLQ-H&N35) | Enrollment, end of radiotherapy (week 7 from start), week 6-8 after the end of radiotherapy, 12, 24, 36, 48, 60 Month after the end of radiotherapy or death from any cause, or last follow-up, whichever occurs first.
  EORTC QLQ-H&N35 quest, specifically tailored for head and neck cancer patients, captures detailed information on a wide range of symptoms and treatment-related toxicities, including but not limited to:
  Dysphagia (difficulty swallowing);Speech problems (articulation and clarity); Xerostomia (dry mouth) Sticky saliva Altered taste and smell Hearing loss Pain in the mouth, throat or jaw Soreness or discomfort in the treated area Breathing difficulties Nasal congestion or discharge Difficulty eating or maintaining weight Nutritional supplementation requirements Body image concerns Social functioning and isolation Financial burden associated with treatment Skin reactions in the irradiated area Fatigue and general physical discomfort Scores for each scale range from 0 to 100. Higher scores on symptom scales indicate worse outcomes (e.g. more pain, worse swallowing), while higher scores on functional scales suggest better outcomes(e.g. improved ability to swallow or speak).
Factors Influencing Recurrence Patterns | From treatment start until first evident recurrence. Censoring for all patients without recurrence at 5 Years.
  Factors Influencing Recurrence Patterns:
  Tumor-Specific Factors:
  Tumor stage and size (T and N classification). Histological subtype and grade. Human papillomavirus (HPV) status: HPV-positive tumors typically have better local and regional control but can still metastasize.
  Treatment-Related Factors:
  Dose and technique of radiotherapy: Modern techniques like IMRT/VMAT with simultaneous integrated boost (SIB) can reduce local recurrence by improving dose conformity.
  Use of concurrent chemotherapy: Enhances radiosensitivity and reduces recurrence risk, especially in advanced-stage disease.
  Adherence to treatment protocols.
  Patient-Specific Factors:
  Smoking and alcohol use post-treatment. Comorbidities that impact treatment tolerance and immune response. Nutritional and functional status.

CONTACTS AND LOCATIONS:
Overall Officials: Victor Lewitzki, MD, PhD, Principal Investigator — University Clinic of Wuerzburg, Department of Radiation Oncology
Locations (1):
- University Clinic of Wuerzburg, Würzburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared publicly due to privacy concerns and ethical considerations. The study ensures strict compliance with data protection regulations, including the anonymization of data stored in a secure, password-protected system within the University Hospital Würzburg's internal network. The sensitive nature of the data, combined with its use for internal quality assurance and prospective analysis, limits its availability for external distribution. Findings and aggregated results will be shared through peer-reviewed publications and presentations, ensuring patient confidentiality is maintained.